CLINICAL TRIAL: NCT05925166
Title: Safety and Efficacy of Of Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ Fusion Protein In Acute Gout
Brief Title: Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ Fusion Protein in the Treatment of Acute Gout
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lihua Duan (Other)
Responsible Party: Sponsor-Investigator, Lihua Duan, Head of rheumatology and immunology, Jiangxi Provincial People's Hopital
Organization: Jiangxi Provincial People's Hopital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DLH86895639
Record Dates: First submitted 2023-06-09; First posted 2023-06-29 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Acute Gout
Keywords: rhTNFR-Fc、Acute Gout
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhTNFR-Fc (Experimental): Subjects will be administered rhTNFR-Fc 50 mg subcutaneously
  Interventions: Drug: rhTNFR-Fc
- Triamcinolone acetonide (Active Comparator): Subjects will be administered triamcinolone acetonide 40 mg intramuscularly
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: rhTNFR-Fc — Subjects will receive 50 mg of study drug on visit 1. A second dose of study drug will be administered if the pain intensity is ≥ 5 on a pain scale of 0-10 at Visit 2
  Other Names: etanercept、Yisaipu
  Arms: rhTNFR-Fc
Drug: Triamcinolone Acetonide — Subjects will be administered triamcinolone acetonide 40 mg intramuscularly on visit 1. A second dose of drug will be administered if the pain intensity is ≥ 5 on a pain scale of 0-10 at Visit 2
  Other Names: Triamcinolone Acetonide Injection
  Arms: Triamcinolone acetonide

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of Recombinant Human Tumor necrosis Factor-α Receptor Ⅱ Fusion Protein （rhTNFR-Fc）in the treatment of patients with acute Gout.

DETAILED DESCRIPTION:
Gout is a disease in which uric acid level exceeds its saturation in blood or tissue fluid due to purine metabolism disorder, excessive production or reduced excretion of uric acid, and thus sodium urate crystals are formed and deposited locally in joints, inducing local inflammatory response and tissue destruction. According to the guidelines for the diagnosis and treatment of gout, it is recommended to use small doses of colchicine or NSAID or glucocorticoid as early as possible (sufficient amount and short course) for treatment in the acute stage of gouty arthritis. Gout patients with intolerance, poor efficacy or contraindications of the above-mentioned drugs are usually considered as refractory gout, which is difficult to treat and lacks universally effective drugs. Recombinant human tumor necrosis factor-α receptor Ⅱ fusion protein（rhTNFR-Fc） has effective anti-inflammatory effect in rheumatoid arthritis, ankylosing spondylitis and other rheumatic diseases. This is a multicenter, prospective, open-label, two-arm study.Subjects will be administered a single dose of rhTNFR-Fc 50 mg subcutaneously (SC), at the onset of an acute gout attack, or a single dose of triamcinolone acetonide 40 mg intramuscularly (IM)，to evaluate the efficacy and safety of rhTNFR-Fc in the treatment of patients with acute Gout.

ELIGIBILITY:
Inclusion Criteria:

1. Can voluntarily sign the informed consent, and voluntarily cooperate with the completion of the experiment according to the plan;
2. 18 years old ≤ 75 years old, male and female;
3. Body mass index (BMI) ≤ 40 kg/m2;
4. Patients diagnosed with gout according to the American College of Rheumatology (ACR) 2015 gout classification criteria;
5. The current acute gout attack occurred within 4 days before the screening period;
6. The pain degree of target joint during the screening period was VAS≥ 5 mm (VAS 0-10mm);
7. We are willing to follow the protocol of uric acid lowering therapy (ULT) during the study period and meet the following conditions One:

(1) Patients who are receiving ULT and stable treatment for ≥14 days should maintain the stable medication regimen for at least 12 weeks during the trial period. Unless the patient with the original uric-lowering regimen is evaluated by the investigator as having intolerance, poor efficacy or low uric acid, adjustment of the uric-lowering regimen including drug change, dose reduction or drug discontinuation is allowed;

② Patients who did not use ULT before randomization were not allowed to take uric-lowering therapy within 14 days after randomization. After 14 days, researchers decided whether to take uric-lowering therapy according to uric acid level. In principle, allopurinol was not used for uric-lowering therapy.

(3) Patients who took ULT before randomization but did not stabilize for 14 days were not allowed to take urico-lowering therapy within 14 days after randomization, and the researchers decided whether to take urico-lowering therapy after 14 days according to the uric acid level. In principle, patients who had not used allopurinol before should not use allopurinol for urico-lowering therapy in this study.

Exclusion Criteria:

1. There is a history of allergic reaction to the investigational drug or similar drugs;
2. People who have received any of the following drugs or treatments:

   1. Use of NASIADs within 24 hours prior to enrollment;
   2. Used ≥ 5 mg prednisone or equivalent dose of glucocorticoid in the 24 hours prior to enrollment;
   3. used short-acting painkillers such as tramadol within 24 hours before enrollment;
   4. Use of long-acting opioid therapy within 14 days prior to screening;
   5. Intraarticular injection of glucocorticoids within 14 days prior to screening;
   6. Use of any IL-1 blocker, TNF inhibitor, or other biologics within 30 days prior to screening or within 3 half-lives, whichever is older;
   7. Continued treatment with systemic immunosuppressive agents for 3 months prior to screening.
3. There are active bleeding diseases of internal organs, or there is a serious bleeding tendency (such as hemophilia, etc.), or anti-coagulation treatment with heparin;
4. Those diagnosed with secondary gout (e.g. chemotherapy-induced gout, lead-induced gout, transplantable gout, etc.Except for gout caused by impaired renal function);
5. Diagnosis or suspicion of rheumatoid arthritis, infectious/septic arthritis, the presence of other conditions that may confuse the assessment of the affected joint, such as the presence of other pain, including but not limited to nerve disease, nerve root compression due to disc herniation, shingles, sciatica, etc.;
6. There are infections requiring systemic drug control within 7 days prior to screening;
7. Have received live or attenuated vaccines within 3 months prior to screening, or plan to receive live or attenuated vaccines during the study period;
8. Those who received COVID-19 vaccine within 2 weeks prior to screening;
9. Cancer within 5 years prior to screening:
10. A history of severe immunodeficiency, including: positive for human immunodeficiency virus (HIV) antibodies; Or other acquired or congenital immunodeficiency diseases;
11. Presence of the following clinically significant diseases:

    1. Patients with a history of chronic congestive heart failure and NYHA level IV cardiac function; Patients with a history of cardiac ejection fraction (EF) less than 30% detected by echocardiography;
    2. Patients with myocardial infarction, acute coronary syndrome, viral myocarditis, or pulmonary embolism within 6 months; Patients who underwent coronary revascularization within 6 months; C. The presence of severe arrhythmias requiring Class Ia or III antiarrhythmic drugs; Arrhythmias with diseased sinus syndrome, grade II type II or grade III atrioventricular block, and no pacemaker implanted;
12. TB T-SPOT or γ interferon release test positive or have a previous history of TB;
13. Hepatitis B surface antigen positive ;
14. Receive kidney dialysis treatment;
15. There are the following abnormalities in the laboratory test values during the screening period:

    1. White blood cell count ≤3×109 /L or neutrophil absolute value ≤1.5×109 /L;
    2. PLT≤100×109 /L;
    3. Total bilirubin >1.5×ULN, alanine aminotransferase (AST) >3×ULN, aspartate aminotransferase (ALT) >;3×ULN;
    4. Estimated glomerular filtration rate (eGFR) < 30ml/min/1.73m2;
16. Pregnant or nursing (lactating) women;
17. Female patients who are biologically capable of becoming pregnant must use an acceptable method of contraception;
18. A history of drug and/or alcohol abuse or mental disorders;
19. It is determined by the investigator that the subject has a history of certain diseases that are not suitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Joint pain intensity in the most affected joint | 72 hours
  Pain intensity in the most affected baseline joint measured by the numeric 0-10 pain scale at 72 hours
Acute gout recurrence time | within 12 weeks
  Time from baseline to first acute gout recurrence

SECONDARY OUTCOMES:
Joint pain on numeric pain scale | Days 4, 7, and 14
  Patient's assessment of joint pain intensity in the most affected baseline joint on a 0-10 pain scale, at Baseline and post-dose Days
Patient's assessment of response to treatment | Day 4, 7 and 14
  Patient's global assessment of response to treatment
Physician's assessment of response to treatment | Day 4, 7 and 14
  Physician's global assessment of response to treatment
Rescue Medication | Days 4, 7, 14
  Compare the use of rescue medication
Safety and Tolerability of rhTNFR-Fc | Days1, 4, 7, 14
  Safety and tolerability as assessed by subjects with adverse events and serious adverse events from baseline through Visit 5 safety follow-up
inflammatory index change | 1week
  Inflammatory index 1 week after treatment: change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lihua Duan, MD, Principal Investigator — Jiangxi Provincial People's Hopital
Locations (1):
- Department of Rheumatology and Clinical Immunology, Jiangxi Provincial People's Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No